CLINICAL TRIAL: NCT02249481
Title: A Comparison of Continuous Adductor Canal Catheter Infusion vs Continuous Femoral Nerve Catheter Infusion for Total Knee Replacement Surgery
Brief Title: A Comparison of Anaesthetic Methods for Total Knee Replacement Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: A number of issues which impact on the ability to recruit patients to the study
Sponsor: University Hospital Plymouth NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14/P/132
Record Dates: First submitted 2014-09-18; First posted 2014-09-25 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-08

CONDITIONS: Total Knee Replacement
Keywords: Anaesthetic; total knee replacement; Femoral nerve catheter; Adductor canal catheter
MeSH Terms: interventions — Levobupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group F (Active Comparator): Femoral nerve catheter delivering 0.0625% L- Bupivacaine: Blockade at level of Femoral crease. Identify femoral nerve. In plane lateral approach. Bolus 20 mls via needle. Catheter threaded and 2-4cm left in situ (bevel orientated cephalad).and 5 mls injected via catheter to confirm spread under ultrasound guidance. Glue/Lockit dressing.
  Interventions: Procedure: Femoral nerve catheter delivering 0.0625% L- Bupivacaine
- Group A (Experimental): Adductor canal catheter delivering 0.0625% L- Bupivacaine: Blockade at mid-thigh. Identify sartorius at mid thigh - find point where the femoral artery begins to descend from sartorius. In plane technique, hydro-dissect space between sartorius and femoral artery. Catheter threaded and 2-4cm left in situ (bevel orientated cephalad). Bolus 20 mls via needle and 5 mls via catheter to confirm spread under ultrasound guidance. Glue/Lockit dressing.
  Interventions: Procedure: Adductor Canal catheter delivering 0.0625% L- Bupivacaine

INTERVENTIONS:
Procedure: Adductor Canal catheter delivering 0.0625% L- Bupivacaine — Adductor canal catheter: Blockade at mid-thigh. Identify sartorius at mid thigh - find point where the femoral artery begins to descend from sartorius. In plane technique, hydro-dissect space between sartorius and femoral artery. Catheter threaded and 2-4cm left in situ (bevel orientated cephalad). Bolus 20 mls via needle and 5 mls via catheter to confirm spread under ultrasound guidance. Glue/Lockit dressing.
  Other Names: Adductor Canal Block (0.0625% L- Bupivacaine)
  Arms: Group A
Procedure: Femoral nerve catheter delivering 0.0625% L- Bupivacaine — Femoral nerve catheter: Blockade at level of Femoral crease. Identify femoral nerve. In plane lateral approach. Bolus 20 mls via needle. Catheter threaded and 2-4cm left in situ (bevel orientated cephalad).and 5 mls injected via catheter to confirm spread under ultrasound guidance. Glue/Lockit dressing.
  Other Names: Femoral nerve Block (0.0625% L- Bupivacaine)
  Arms: Group F

SUMMARY:
Open-labelled, randomised controlled trial. Patients will be assessed pre-operatively, at 24 and 48 hours for the primary outcome and secondary outcomes (except for Oxford Knee Score which will be assessed pre-operatively and at 6 months post-operatively by the ortho-paedic team).

Primary Objective: To demonstrate whether adductor canal nerve infusions result in superior patient mobilisation within the first 48 hours following total knee replacement compared to femoral nerve catheter infusions.

Secondary Objective: To identify whether adductor canal nerve infusions result in superior analgesia within the first 48 hours following total knee replacement compared to femoral nerve catheter infusions.

DETAILED DESCRIPTION:
We are comparing a continuous adductor canal block with a low concentration continuous femoral nerve block. We currently use a low dose femoral nerve catheter based technique as part of our standard treatment strategy for total knee arthroplasty. The use of a catheter provides prolonged analgesia compared to a single shot block, and also allows a lower concentration of local anaesthetic to be employed, thus potentially reducing the incidence of motor blockade. The concentration of local anaesthetic employed in our routine practice (0.0625% L- Bupivacaine) is lower than that routinely used in many other centres, and most clinical studies have compared higher concentrations of local anaesthetic - this might be expected to produce more motor blockade. The concentration we use is higher than the minimum effective concentration for a femoral catheter infusion for knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a diagnosis of rheumatoid or osteoarthritis and listed for a primary total knee replacement.
* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged between 18 and 85 years.
* American Society of Anesthesiologists (ASA) score I-III
* Able (in the clinical staff's opinion) and willing to comply with all study requirements.
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be noti-fied of participation in the study.

Exclusion Criteria:

* Patient refusal
* Chronic pain (defined as consumption of >480mg codeine/24hrs or ANY regular strong opiate consumption by the oral/transdermal route)
* Patients aged <18 or >85
* ASA score >III
* Body mass index (BMI) >35
* Lacking mental capacity to give consent to enter trial/undergo surgery
* Contraindications to catheter placement (coagulopathy , systemic sepsis or infection at placement site, pre-existing neuropathy) or any other component to the study treatment pathway.
* Participant who is terminally ill
* Allergy/intolerance to study medications
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-12-08 (Actual); Primary Completion 2017-06-27 (Actual); Study Completion 2017-06-27 (Actual)

PRIMARY OUTCOMES:
Timed Up Go (TUG) test | 24 hours post-op
  This measures the time (in seconds) taken by a patient to rise to their feet from a sitting position, walk 3 metres in a straight line, turn around, walk back to the seat and sit down again.
Timed Up Go (TUG) test | 48 hours post-op
  This measures the time (in seconds) taken by a patient to rise to their feet from a sitting position, walk 3 metres in a straight line, turn around, walk back to the seat and sit down again.

SECONDARY OUTCOMES:
Total opiate consumption | 48 hours post-op
  morphine equivalence
Visual Analogue Score (VAS) for pain | 24 and 48 hours post-op
  Both at rest and on active movement
Range of knee flexion | 24 and 48 hours post-op
  The range of flexion movement (in degrees) is recorded using a goniometer
Maximum Voluntary Isometric Contraction (MVIC) | 24 and 48 hours post-op
  The quadriceps muscle power in the operative leg is assessed using a handheld dynamometer (HHD)
Oxford Knee Score (OKS) | Pre-op, and at 6 months post-op
  Patient reported outcome score.

CONTACTS AND LOCATIONS:
Overall Officials: Matt Oldman, MB BS, FRCA, Principal Investigator — University Hospital Plymouth NHS Trust
Locations (1):
- Plymouth Hospitals NHS Trust, Plymouth, Devon, United Kingdom